CLINICAL TRIAL: NCT03994445
Title: Effectiveness of Mobile Phone-Based Intervention to Prevent Smoking Relapse Among Recent Smoking Quitters in Jazan Region: Randomized Control Trial.
Brief Title: Effectiveness of Mobile Phone-Based Intervention to Prevent Smoking Relapse Among Recent Smoking Quitters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ibtihal Altalhi (Other)
Responsible Party: Sponsor-Investigator, Ibtihal Altalhi, Dr, King Khalid University
Organization: King Khalid University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SRP in recently quit smokers
Record Dates: First submitted 2019-06-12; First posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group will be enrolled to the intervention program proposed to be (pharmacotherapy + counseling+ motivator phone messages).
  Interventions: Behavioral: Mobile Phone-Based Intervention
- Control group (No Intervention): Control group will receive the standard treatment of the Ministry of the Health program (pharmacotherapy + counseling) only.

INTERVENTIONS:
Behavioral: Mobile Phone-Based Intervention — We propose our intervention based on social cognitive behavior theories and the stages of the change model.
  The program will be carried out using the word "Mettle", it will help ex-smokers stay off cigarettes through advices generated to promote the health from religious concepts and culture perspectives .
  Arms: Intervention group

SUMMARY:
Main Objective The main objective of the study is to investigate the effectiveness of a mobile phone-based intervention in reducing relapse ate among recent quitters who are attending the smoking cessation program in Jazan.

Besides this, the study will achieve the following objective:

To identify the timing and different factors associated with relapse process among recent quitters during first 6 months of quitting.

DETAILED DESCRIPTION:
Background:

Smoking remains a major public health problem and an important cause of morbidity and mortality worldwide. Although the effectiveness of behavior support and medical treatment, many of those who quit smoking subsequently relapse to smoke.

Objective:

The primary aim of this study will be to determine the effectiveness of the mobile phone-based intervention to prevent relapse among recent smoking quitters. Also, the study aims to identify the different factors associated with relapse among recent quitters during the first 6 months of quitting.

Design and Methods:

A parallel two-armed Randomized Controlled Trial (RCT) to assess the effectiveness of a mobile phone-based intervention for smoking cessation on achieving long term abstinence, will be conducted among volunteers. Participants will be recruited from those attended smoking cessation program in Southern Alrawdha clinic, Southern Abo Arish clinic, Sabia clinic and Aldhabia clinic.

Primary outcome:

The difference in relapsing rate among recent quitters, which may subsequently contribute in to a reduction in smoking rates.

Trail Implications for public Health:

The result of this study will provide evidence for effectiveness of the mobile phone-based intervention versus standard treatment to reduce smoking relapse rate. If proven, it will be a cost-saving intervention by reducing repeat use of the smoking cessation clinic services and by reducing use of healthcare services for smoking-related illness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Recent quitters (24 hours smoking abstinence)
* Willing to provide informed consent to participate in the study.

Exclusion Criteria:

* Those suffering any physical or mental disorders.
* Illiterate people.
* Pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
The primary study outcome will be the difference at 6 months relapse rate between the two arms, relapse rate will be identified as a return to continuous smoking even a puff after obtaining 24 hours of abstinence | 6 months following scheduled quit date
  Relapse rates at the end of the 3rd and 6th month of follow-up in the intervention and control groups.

SECONDARY OUTCOMES:
Secondary outcomes included: (1) timing till self-reported relapse. (2) causes of relapse. | 6 months following scheduled quit date
  Participants will be asked core smoking status questions, including whether they have smoked any cigarettes or used other tobacco products, even a puff, in the last 30 days, 7-day point prevalence abstinence, the exact day of each smoking relapse episode and the cause of relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Mahfouz, ASSC PROF, Study Director — University of Jazan
Locations (1):
- Smoking Cessation Clinic - Ministry of Health, Jizan, Saudi Arabia